CLINICAL TRIAL: NCT01905033
Title: Molecular Diagnosis and Risk Stratification of Sepsis
Acronym: MARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Center for Translational Molecular Medicine (Other); UMC Utrecht (Other); Radboud University Medical Center (Other); Philips Healthcare (Industry); Microbiome (Unknown); Immunetrics (Unknown); Check-Points (Unknown); Biocartis NV (Industry); Immunexpress (Industry)
Responsible Party: Principal Investigator, T. van der Poll, Prof. dr. T. van der Poll, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 10-056
Record Dates: First submitted 2013-07-11; First posted 2013-07-23 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Sepsis
Keywords: Sepsis; Pneumonia; Peritonitis; Biomarkers; Transcriptomics; Pathogen detection
MeSH Terms: conditions — Sepsis; Pneumonia; Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood, plasma, RNA, DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Sepsis is a major cause of in-hospital morbidity and mortality. Current tools available to the clinician to initiate therapy of patients with sepsis mainly comprise of symptom classification systems and culture techniques, which provide aspecific and slow information.

Objective: The ultimate goal of this program is to assist the physician at the bedside in tailoring the treatment of an individual patient suffering from sepsis by generating rapid molecular information about the causative pathogen and the host response.

Deliverables: Rapid tests ("sample-in-result-out") that can be used by health care personnel at or close to the bedside and that provide rapid information (within two hours) about the presence or absence of sepsis, the causative pathogen and the risk of the individual patient for sepsis complications and death.

Design: The program is organized into four Work Packages (WPs) along a clinical, discovery and technology platform. In WP1 two university hospitals will enroll 7500 patients admitted to the Intensive Care Unit during the first 3 years of the project; 25% - 40% of these patients will have or will develop sepsis. In WP2 (Pathogen Detection), blood obtained from these patients will be used to develop rapid, fully automated DNA-based bedside tests that identify microorganisms and also provide information about their resistance to antibiotics. In WP3 (Host Response), RNA from blood cells will be analyzed to find novel biomarkers and to develop rapid and easy to perform tests that provide information about the risk profile of the patient. In addition, plasma levels of selected protein biomarkers will be measured for comparison of their value with that of the identified leukocyte molecular signatures. WP4 is responsible for the ICT management of the project. The Clinical Platform (covered by WP1 and WP4) delivers patient data and biological samples to the discovery and technology platforms. The Discovery Platform (covered by WP2 and WP3) uses patient data and biological samples to develop tests for detection of the infectious agent causing sepsis and for stratification of patients according to their risk for sepsis complications, including death. The results generated within the discovery platform will be delivered to the technology platform. The Technology Platform (part of WP2 and WP3) has the specific aim to develop rapid assays that run on a fully automated (micro)fluidics platform that is so easy to operate that it can be used in decentralized settings such as (close to) the ICU. The developed assays will make use of the knowledge generated in the discovery platform.

ELIGIBILITY:
Inclusion Criteria:

* All patients> 18 years in the Intensive Care Units of the AMC Amsterdam and UMC Utrecht.

Exclusion Criteria:

* Elective cardiac surgery patients with an uncomplicated stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 3-4 years all patients> 18 years in the Intensive Care Units of the AMC Amsterdam and UMC Utrecht will be included in the study with the exemption of elective cardiac surgery patients with an uncomplicated stay.
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Molecular information about causative pathogens and the host response in patients with sepsis | One year

SECONDARY OUTCOMES:
Stratification of septic patients by severity and type of immune response to infection | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Tom van der Poll, Prof., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam, North Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

REFERENCES:
- [Derived] Scicluna BP, Cano-Gamez K, Burnham KL, Davenport EE, Moore AR, Khan S, Hinds CJ, Cremer OL, Khatri P, Sweeney TE, Knight JC, van der Poll T. A consensus blood transcriptomic framework for sepsis. Nat Med. 2025 Dec;31(12):4119-4130. doi: 10.1038/s41591-025-03964-5. Epub 2025 Sep 30. PMID 41028542
- [Derived] Filippini DFL, Jiang M, Kramer L, van der Poll T, Cremer O, Hla TTW, Retter A, Bos LDJ; MARS consortium. Plasma H3.1 nucleosomes as biomarkers of infection, inflammation and organ failure. Crit Care. 2025 May 19;29(1):198. doi: 10.1186/s13054-025-05415-6. PMID 40390092
- [Derived] Brands X, Uhel F, van Vught LA, Wiewel MA, Hoogendijk AJ, Lutter R, Schultz MJ, Scicluna BP, van der Poll T. Immune suppression is associated with enhanced systemic inflammatory, endothelial and procoagulant responses in critically ill patients. PLoS One. 2022 Jul 25;17(7):e0271637. doi: 10.1371/journal.pone.0271637. eCollection 2022. PMID 35877767
- [Derived] Peters-Sengers H, Butler JM, Uhel F, Schultz MJ, Bonten MJ, Cremer OL, Scicluna BP, van Vught LA, van der Poll T; MARS consortium. Source-specific host response and outcomes in critically ill patients with sepsis: a prospective cohort study. Intensive Care Med. 2022 Jan;48(1):92-102. doi: 10.1007/s00134-021-06574-0. Epub 2021 Dec 13. PMID 34902047
- [Derived] Frencken JF, van Smeden M, van de Groep K, Ong DSY, Klein Klouwenberg PMC, Juffermans N, Bonten MJM, van der Poll T, Cremer OL; MARS Consortium. Etiology of Myocardial Injury in Critically Ill Patients with Sepsis: A Cohort Study. Ann Am Thorac Soc. 2022 May;19(5):773-780. doi: 10.1513/AnnalsATS.202106-689OC. PMID 34784496
- [Derived] Pereverzeva L, Uhel F, Peters Sengers H, Cremer OL, Schultz MJ, Bonten MMJ, Scicluna BP, van der Poll T; MARS consortium. Association between delay in intensive care unit admission and the host response in patients with community-acquired pneumonia. Ann Intensive Care. 2021 Sep 28;11(1):142. doi: 10.1186/s13613-021-00930-5. PMID 34585271
- [Derived] Brands X, de Vries FMC, Uhel F, Haak BW, Peters-Sengers H, Schuurman AR, van Engelen TSR, Lutter R, Cremer OL, Bonten MJ, Schultz MJ, Scicluna BP, van der Poll T; MARS Consortium. Plasma Ferritin as Marker of Macrophage Activation-Like Syndrome in Critically Ill Patients With Community-Acquired Pneumonia. Crit Care Med. 2021 Nov 1;49(11):1901-1911. doi: 10.1097/CCM.0000000000005072. PMID 33935163
- [Derived] Simonis FD, Schouten LRA, Cremer OL, Ong DSY, Amoruso G, Cinella G, Schultz MJ, Bos LD; MARS consortium. Prognostic classification based on P/F and PEEP in invasively ventilated ICU patients with hypoxemia-insights from the MARS study. Intensive Care Med Exp. 2020 Dec 18;8(Suppl 1):43. doi: 10.1186/s40635-020-00334-y. PMID 33336322
- [Derived] Uhel F, Peters-Sengers H, Falahi F, Scicluna BP, van Vught LA, Bonten MJ, Cremer OL, Schultz MJ, van der Poll T; MARS consortium. Mortality and host response aberrations associated with transient and persistent acute kidney injury in critically ill patients with sepsis: a prospective cohort study. Intensive Care Med. 2020 Aug;46(8):1576-1589. doi: 10.1007/s00134-020-06119-x. Epub 2020 Jun 8. PMID 32514599
- [Derived] Klein Klouwenberg PMC, Spitoni C, van der Poll T, Bonten MJ, Cremer OL; MARS consortium. Predicting the clinical trajectory in critically ill patients with sepsis: a cohort study. Crit Care. 2019 Dec 12;23(1):408. doi: 10.1186/s13054-019-2687-z. PMID 31831072
- [Derived] Schouten LRA, Bos LDJ, Serpa Neto A, van Vught LA, Wiewel MA, Hoogendijk AJ, Bonten MJM, Cremer OL, Horn J, van der Poll T, Schultz MJ, Wosten-van Asperen RM; MARS consortium. Increased mortality in elderly patients with acute respiratory distress syndrome is not explained by host response. Intensive Care Med Exp. 2019 Oct 29;7(1):58. doi: 10.1186/s40635-019-0270-1. PMID 31664603
- [Derived] Verboom DM, Frencken JF, Ong DSY, Horn J, van der Poll T, Bonten MJM, Cremer OL, Klein Klouwenberg PMC. Robustness of sepsis-3 criteria in critically ill patients. J Intensive Care. 2019 Aug 29;7:46. doi: 10.1186/s40560-019-0400-6. eCollection 2019. PMID 31489199
- [Derived] Frencken JF, van Baal L, Kappen TH, Donker DW, Horn J, van der Poll T, van Klei WA, Bonten MJM, Cremer OL; Members of the MARS Consortium. Myocardial Injury in Critically Ill Patients with Community-acquired Pneumonia. A Cohort Study. Ann Am Thorac Soc. 2019 May;16(5):606-612. doi: 10.1513/AnnalsATS.201804-286OC. PMID 30521759
- [Derived] Miller RR 3rd, Lopansri BK, Burke JP, Levy M, Opal S, Rothman RE, D'Alessio FR, Sidhaye VK, Aggarwal NR, Balk R, Greenberg JA, Yoder M, Patel G, Gilbert E, Afshar M, Parada JP, Martin GS, Esper AM, Kempker JA, Narasimhan M, Tsegaye A, Hahn S, Mayo P, van der Poll T, Schultz MJ, Scicluna BP, Klein Klouwenberg P, Rapisarda A, Seldon TA, McHugh LC, Yager TD, Cermelli S, Sampson D, Rothwell V, Newman R, Bhide S, Fox BA, Kirk JT, Navalkar K, Davis RF, Brandon RA, Brandon RB. Validation of a Host Response Assay, SeptiCyte LAB, for Discriminating Sepsis from Systemic Inflammatory Response Syndrome in the ICU. Am J Respir Crit Care Med. 2018 Oct 1;198(7):903-913. doi: 10.1164/rccm.201712-2472OC. PMID 29624409
- [Derived] Cranendonk DR, van Vught LA, Wiewel MA, Cremer OL, Horn J, Bonten MJ, Schultz MJ, van der Poll T, Wiersinga WJ. Clinical Characteristics and Outcomes of Patients With Cellulitis Requiring Intensive Care. JAMA Dermatol. 2017 Jun 1;153(6):578-582. doi: 10.1001/jamadermatol.2017.0159. PMID 28296993
- [Derived] Ong DSY, Bonten MJM, Spitoni C, Verduyn Lunel FM, Frencken JF, Horn J, Schultz MJ, van der Poll T, Klein Klouwenberg PMC, Cremer OL; Molecular Diagnosis and Risk Stratification of Sepsis Consortium. Epidemiology of Multiple Herpes Viremia in Previously Immunocompetent Patients With Septic Shock. Clin Infect Dis. 2017 May 1;64(9):1204-1210. doi: 10.1093/cid/cix120. PMID 28158551
- [Derived] Wiewel MA, Harmon MB, van Vught LA, Scicluna BP, Hoogendijk AJ, Horn J, Zwinderman AH, Cremer OL, Bonten MJ, Schultz MJ, van der Poll T, Juffermans NP, Wiersinga WJ. Risk factors, host response and outcome of hypothermic sepsis. Crit Care. 2016 Oct 14;20(1):328. doi: 10.1186/s13054-016-1510-3. PMID 27737683
- [Derived] Klein Klouwenberg PM, Frencken JF, Kuipers S, Ong DS, Peelen LM, van Vught LA, Schultz MJ, van der Poll T, Bonten MJ, Cremer OL; MARS Consortium *. Incidence, Predictors, and Outcomes of New-Onset Atrial Fibrillation in Critically Ill Patients with Sepsis. A Cohort Study. Am J Respir Crit Care Med. 2017 Jan 15;195(2):205-211. doi: 10.1164/rccm.201603-0618OC. PMID 27467907
- [Derived] McHugh L, Seldon TA, Brandon RA, Kirk JT, Rapisarda A, Sutherland AJ, Presneill JJ, Venter DJ, Lipman J, Thomas MR, Klein Klouwenberg PM, van Vught L, Scicluna B, Bonten M, Cremer OL, Schultz MJ, van der Poll T, Yager TD, Brandon RB. A Molecular Host Response Assay to Discriminate Between Sepsis and Infection-Negative Systemic Inflammation in Critically Ill Patients: Discovery and Validation in Independent Cohorts. PLoS Med. 2015 Dec 8;12(12):e1001916. doi: 10.1371/journal.pmed.1001916. eCollection 2015 Dec. PMID 26645559
- [Derived] Klein Klouwenberg PM, Cremer OL, van Vught LA, Ong DS, Frencken JF, Schultz MJ, Bonten MJ, van der Poll T. Likelihood of infection in patients with presumed sepsis at the time of intensive care unit admission: a cohort study. Crit Care. 2015 Sep 7;19(1):319. doi: 10.1186/s13054-015-1035-1. PMID 26346055
- [Derived] Scicluna BP, Klein Klouwenberg PM, van Vught LA, Wiewel MA, Ong DS, Zwinderman AH, Franitza M, Toliat MR, Nurnberg P, Hoogendijk AJ, Horn J, Cremer OL, Schultz MJ, Bonten MJ, van der Poll T. A molecular biomarker to diagnose community-acquired pneumonia on intensive care unit admission. Am J Respir Crit Care Med. 2015 Oct 1;192(7):826-35. doi: 10.1164/rccm.201502-0355OC. PMID 26121490
- [Derived] Klein Klouwenberg PM, Zaal IJ, Spitoni C, Ong DS, van der Kooi AW, Bonten MJ, Slooter AJ, Cremer OL. The attributable mortality of delirium in critically ill patients: prospective cohort study. BMJ. 2014 Nov 24;349:g6652. doi: 10.1136/bmj.g6652. PMID 25422275